CLINICAL TRIAL: NCT03371199
Title: The Effect of Normalization of Sodium on Bone Markers in Patients With Epilepsy. A Randomized Single-blinded Placebo-controlled Trial.
Brief Title: The Association Between Hyponatremia and Osteoporosis in Patients With Epilepsy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Sarah Seberg Diemar, Medical Doctor, ph.d. student, principal investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 57353
Record Dates: First submitted 2017-11-30; First posted 2017-12-13 (Actual); Last update posted 2019-03-28 (Actual); Status verified 2019-03

CONDITIONS: Hyponatremia; Metabolic Bone Disease
MeSH Terms: conditions — Hyponatremia; Bone Diseases, Metabolic | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sodium arm (Active Comparator): Sodium tablets
  Interventions: Drug: Sodium chloride
- Placebo arm (Placebo Comparator): Placebo tablets
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Sodium chloride — Sodium chloride tablets, 250 mg
  Arms: Sodium arm
Drug: Placebo Oral Tablet — Starch tablets
  Other Names: Strarch tablets
  Arms: Placebo arm

SUMMARY:
The study investigates the association between normalization of serum sodium levels and bone markers in patients with epilepsy and chronic hyponatremia.

The study is a randomized, single blinded, placebo controlled study where participants will be randomized to either treatment with salt tablets or placebo tablets through 4 months. At the beginning and end of the 4 months bone markers will be measured.

The investigators null-hypothesis is that there will be no difference in bone markers before or after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Epilepsy requiring treatment for at least 2 years
* Known hyponatremia (2 subsequent s-sodium values < 136 mmol/l)
* Age 18-80 years
* Danish speaking
* Signed form of prior consent

Exclusion Criteria:

* Pregnancy and breastfeeding
* Known osteoporosis. DXA scan < -2.5 T-score. Z-score is used for patients 50 years or younger.
* Undergoing treatment for osteoporosis
* Undergoing treatment with salt tablets
* Known SIADH
* Severe concomitant disease such as cancer or ischemic heart disease
* Alcohol, drug or substance abuse

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
CTX1 change | At baseline and after 4 months intervention
  bone markers

SECONDARY OUTCOMES:
P1NP change | At baseline and after 4 months intervention
  Bone markers
DXA scan change | At baseline and after 4 months intervention
  Density measurements
Cognitive function change | At baseline and after 4 months intervention
  Epitrack test, scale from 9-49 (9 worst score - 49 best score)
Life quality change | At baseline and after 4 months intervention
  Quoli 31, scale from 0-100 (0 lowest life quality - 100 best life quality)
Change in daily pains | At baseline and after 4 months intervention
  VAS from 0-10 (0 no pains - 10 maximum pain)

CONTACTS AND LOCATIONS:
Overall Officials: Noémi B Andersen, DMSc, MD, Study Chair — Senoir consultant
Locations (1):
- Rigshospitalet Glostrup, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: No
We have currently no plan to share individual patient data, but if relevant if relevant it could occur.

REFERENCES:
- [Background] Fedorenko M, Wagner ML, Wu BY. Survey of risk factors for osteoporosis and osteoprotective behaviors among patients with epilepsy. Epilepsy Behav. 2015 Apr;45:217-22. doi: 10.1016/j.yebeh.2015.01.021. Epub 2015 Mar 24. PMID 25812937
- [Background] Maraka S, Kennel KA. Bisphosphonates for the prevention and treatment of osteoporosis. BMJ. 2015 Sep 2;351:h3783. doi: 10.1136/bmj.h3783. PMID 26333528
- [Background] Darba J, Kaskens L, Perez-Alvarez N, Palacios S, Neyro JL, Rejas J. Disability-adjusted-life-years losses in postmenopausal women with osteoporosis: a burden of illness study. BMC Public Health. 2015 Apr 2;15:324. doi: 10.1186/s12889-015-1684-7. PMID 25880810
- [Background] Wu FJ, Sheu SY, Lin HC. Osteoporosis is associated with antiepileptic drugs: a population-based study. Epileptic Disord. 2014 Sep;16(3):333-42. doi: 10.1684/epd.2014.0673. PMID 25166266
- [Background] Asconape JJ. Some common issues in the use of antiepileptic drugs. Semin Neurol. 2002 Mar;22(1):27-39. doi: 10.1055/s-2002-33046. PMID 12170391
- [Background] Vasikaran S, Eastell R, Bruyere O, Foldes AJ, Garnero P, Griesmacher A, McClung M, Morris HA, Silverman S, Trenti T, Wahl DA, Cooper C, Kanis JA; IOF-IFCC Bone Marker Standards Working Group. Markers of bone turnover for the prediction of fracture risk and monitoring of osteoporosis treatment: a need for international reference standards. Osteoporos Int. 2011 Feb;22(2):391-420. doi: 10.1007/s00198-010-1501-1. Epub 2010 Dec 24. PMID 21184054
- [Background] Sejling AS, Thorsteinsson AL, Pedersen-Bjergaard U, Eiken P. Recovery from SIADH-associated osteoporosis: a case report. J Clin Endocrinol Metab. 2014 Oct;99(10):3527-30. doi: 10.1210/jc.2014-1572. Epub 2014 Jun 27. PMID 24971663
- [Background] Sejling AS, Pedersen-Bjergaard U, Eiken P. Syndrome of inappropriate ADH secretion and severe osteoporosis. J Clin Endocrinol Metab. 2012 Dec;97(12):4306-10. doi: 10.1210/jc.2012-2031. Epub 2012 Oct 17. PMID 23076350
- [Background] Verbalis JG, Barsony J, Sugimura Y, Tian Y, Adams DJ, Carter EA, Resnick HE. Hyponatremia-induced osteoporosis. J Bone Miner Res. 2010 Mar;25(3):554-63. doi: 10.1359/jbmr.090827. PMID 19751154
- [Background] Barsony J, Sugimura Y, Verbalis JG. Osteoclast response to low extracellular sodium and the mechanism of hyponatremia-induced bone loss. J Biol Chem. 2011 Mar 25;286(12):10864-75. doi: 10.1074/jbc.M110.155002. Epub 2010 Dec 6. PMID 21135109
- [Background] Himmerkus N, Sievers B, Bleich M. Carbamazepine affects water and electrolyte homoeostasis in rat--similarities and differences to vasopressin antagonism. Nephrol Dial Transplant. 2012 Oct;27(10):3790-8. doi: 10.1093/ndt/gfs107. Epub 2012 May 4. PMID 22561584